CLINICAL TRIAL: NCT00128700
Title: Phase I/II Study on Concomitant and Adjuvant Temozolomide and Radiotherapy With or Without PTK787/ZK222584 in Newly Diagnosed GBM
Brief Title: Temozolomide and Radiation Therapy With or Without Vatalanib in Treating Patients With Newly Diagnosed Glioblastoma Multiforme
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: European Organisation for Research and Treatment of Cancer - EORTC (Network)
Responsible Party: Sponsor
Allocation: Randomized | Masking: None | Purpose: Treatment
Other Study IDs: EORTC-26041-22041; EORTC-26041; EORTC-22041; EUDRACT-2004-003896-35
Record Dates: First submitted 2005-08-08; First posted 2005-08-10 (Estimated); Last update posted 2012-09-24 (Estimated); Status verified 2012-09

CONDITIONS: Brain and Central Nervous System Tumors
Keywords: adult glioblastoma; adult giant cell glioblastoma; adult gliosarcoma
MeSH Terms: conditions — Central Nervous System Neoplasms; Glioblastoma; Gliosarcoma | interventions — Temozolomide; vatalanib; Chemotherapy, Adjuvant; Radiotherapy

INTERVENTIONS:
Drug: temozolomide
Drug: vatalanib
Procedure: adjuvant therapy
Radiation: radiation therapy

SUMMARY:
RATIONALE: Drugs used in chemotherapy, such as temozolomide, work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing. Radiation therapy uses high-energy x-rays to kill tumor cells. Vatalanib may stop the growth of tumor cells by blocking blood flow to the tumor. Giving temozolomide and radiation therapy together with vatalanib may kill more tumor cells.

PURPOSE: This randomized phase I/II trial is studying the side effects and best dose of vatalanib when given together with temozolomide and radiation therapy and to see how well they work in treating patients with newly diagnosed glioblastoma multiforme.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Determine the maximum tolerated dose and recommended phase II dose of vatalanib when given in combination with temozolomide and radiotherapy in patients with newly diagnosed glioblastoma multiforme. (Phase I)
* Determine the safety and tolerability of this regimen in these patients. (Phase I)
* Determine the 6-month progression-free survival of patients treated with chemoradiotherapy comprising temozolomide and radiotherapy with or without vatalanib followed by adjuvant therapy comprising temozolomide and vatalanib or temozolomide alone with or without maintenance therapy comprising vatalanib alone. (Phase II)

Secondary

* Determine 12-month overall survival of patients treated with these regimens. (Phase II)
* Determine the toxicity profile of these regimens in these patients. (Phase II)
* Correlate expression of angiogenesis and hypoxia markers and MGMT methylation status with clinical outcome in patients treated with these regimens.

OUTLINE: This is a phase I, multicenter, open-label, non-randomized, dose-escalation study of vatalanib followed by a phase II, randomized, controlled study. Patients enrolled in the phase II portion of the study are stratified according to participating center, age (< 50 years vs ≥ 50 years), corticosteroid intake (yes vs no), and mini-mental status evaluation score (< 27 vs 27-29 vs 30).

* Phase I:

  * Chemoradiotherapy: Patients receive oral temozolomide once daily for 6-7 weeks and oral vatalanib once daily for 6 weeks. Patients also undergo radiotherapy once daily, 5 days a week, for 6 weeks. Four weeks after the completion of chemoradiotherapy, patients proceed to adjuvant therapy. During the 4-week period between chemoradiotherapy and adjuvant therapy, patients continue to receive oral vatalanib twice daily.

Cohorts of 3-6 patients receive escalating doses of vatalanib during chemoradiotherapy until the maximum tolerated dose is determined (MTD). The MTD is defined as the dose preceding that at which 2 of 3 or 2 of 6 patients experience dose-limiting toxicity. At least 6 patients are treated at the MTD.

* Adjuvant therapy: Patients receive oral temozolomide once daily on days 1-5 and oral vatalanib twice daily on days 1-28. Treatment repeats every 28 days for 6 courses in the absence of disease progression or unacceptable toxicity. Patients then proceed to maintenance therapy.
* Maintenance therapy: Patients continue to receive oral vatalanib twice daily in the absence of disease progression or unacceptable toxicity.

  * Phase II: Patients are randomized to 1 of 3 treatment arms.
* Arm I:

  * Chemoradiotherapy: Patients receive oral temozolomide once daily for 6-7 weeks and undergo radiotherapy once daily, 5 days a week, for 6 weeks. Four weeks after the completion of chemoradiotherapy, patients proceed to adjuvant therapy.
  * Adjuvant therapy: Patients receive oral temozolomide once daily on days 1-5. Treatment repeats every 28 days for up to 6 courses in the absence of disease progression or unacceptable toxicity.
* Arm II:

  * Chemoradiotherapy: Patients receive temozolomide and undergo radiotherapy as in arm I. Patients also receive vatalanib twice daily for 6 weeks at the MTD determined in phase I. Four weeks after the completion of chemoradiotherapy, patients proceed to adjuvant therapy. During the 4-week period between chemoradiotherapy and adjuvant therapy, patients continue to receive oral vatalanib twice daily.
  * Adjuvant therapy: Patients receive temozolomide and vatalanib as in phase I adjuvant therapy. Patients then proceed to maintenance therapy.
  * Maintenance therapy: Patients continue to receive vatalanib as in phase I maintenance therapy.
* Arm III:

  * Chemoradiotherapy: Patients receive temozolomide and undergo radiotherapy as in arm I. Four weeks after the completion of chemoradiotherapy, patients proceed to adjuvant therapy. During the 4-week period between chemoradiotherapy and adjuvant therapy, patients receive oral vatalanib twice daily.
  * Adjuvant therapy: Patients receive temozolomide and vatalanib as in phase I adjuvant therapy. Patients then proceed to maintenance therapy.
  * Maintenance therapy: Patients continue to receive vatalanib as in phase I maintenance therapy.

After completion of study treatment, patients are followed every 3 months for survival.

PROJECTED ACCRUAL: Approximately 3-18 patients will be accrued for the phase I portion of this study. A total of 201 patients (67 per treatment arm) will be accrued for the phase II portion of this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed glioblastoma multiforme

  * Newly diagnosed disease
* Deemed to be amenable to concurrent and adjuvant temozolomide treatment by the principal investigator

PATIENT CHARACTERISTICS:

Age

* 18 to 69

Performance status

* ECOG 0-1

Life expectancy

* Not specified

Hematopoietic

* Absolute neutrophil count ≥ 1,500/mm^3
* Platelet count ≥ 100,000/mm^3

Hepatic

* Bilirubin < 1.5 times upper limit of normal (ULN)
* Alkaline phosphatase < 2.5 times ULN
* ALT and AST < 2.5 times ULN

Renal

* Creatinine ≤ 1.7 mg/dL

Cardiovascular

* Cardiac function clinically normal
* 12-lead ECG normal
* No ischemic heart disease within the past 6 months
* No uncontrolled cardiac arrhythmia
* No uncontrolled hypertension
* No history of stroke
* No history of congenital long QT syndrome
* QTc interval ≤ 450 msec for males or ≤ 470 msec for females by 12-lead ECG

Other

* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception
* No other malignancy except adequately treated basal cell or squamous cell skin cancer or cone biopsied carcinoma in situ of the cervix
* No active uncontrolled infection
* No other unstable systemic disease
* No psychological, familial, sociological, or geographical condition that would preclude study compliance or follow-up schedule

PRIOR CONCURRENT THERAPY:

Biologic therapy

* No prior anti-vascular endothelial growth factor therapy

Chemotherapy

* No prior chemotherapy

Endocrine therapy

* Concurrent corticosteroids allowed provided the patient is on stable or decreasing doses for ≥ 2 weeks before study entry

Radiotherapy

* No prior radiotherapy

Surgery

* More than 8 days, but < 6 weeks, since prior surgery or biopsy

Other

* No prior randomization on this study
* No concurrent warfarin, warfarin-derived drugs, or similar anticoagulants
* No other concurrent anticancer therapy
* No other concurrent investigational agents
* No concurrent enzyme inducing antiepileptic drugs, including any of the following:

  * Carbamazepine
  * Fosphenytoin
  * Oxcarbazepine
  * Phenobarbital
  * Phenytoin
  * Primidone
* No concurrent grapefruit or grapefruit juice

Ages: 18 Years to 69 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2005-06; Primary Completion 2007-11 (Actual)

PRIMARY OUTCOMES:
Dose-limiting toxicity and maximum tolerated dose of vatalanib as determined by CTCAE v3.0 during phase I
Progression-free survival at 6 months during phase II

SECONDARY OUTCOMES:
Severe toxic events as assessed by CTCAE v3.0 at weeks 3 and 6 (concomitant treatment), weeks 2 and 4 after radiotherapy, before each course of adjuvant treatment, monthly during maintenance treatment, and every 3 months during follow-up in phase II
Overall survival at 1 year during phase II
Correlation of angiogenesis and hypoxia markers expression and O-6-methylguanine DNA methyltransferase (MGMT) methylation status with clinical outcome during phase II

CONTACTS AND LOCATIONS:
Overall Officials: Alba A. Brandes, MD, Study Chair — Azienda Ospedaliera di Padova
Locations (5):
- U.Z. Gasthuisberg, Leuven, Belgium
- Klinikum der Universitaet Regensburg, Regensburg, Germany
- Azienda Ospedaliera di Padova, Padua, Italy
- Daniel Den Hoed Cancer Center at Erasmus Medical Center, Rotterdam, Netherlands
- Centre Hospitalier Universitaire Vaudois, Lausanne, Switzerland

REFERENCES:
- [Result] Brandes AA, Stupp R, Hau P, Lacombe D, Gorlia T, Tosoni A, Mirimanoff RO, Kros JM, van den Bent MJ. EORTC study 26041-22041: phase I/II study on concomitant and adjuvant temozolomide (TMZ) and radiotherapy (RT) with PTK787/ZK222584 (PTK/ZK) in newly diagnosed glioblastoma. Eur J Cancer. 2010 Jan;46(2):348-54. doi: 10.1016/j.ejca.2009.10.029. Epub 2009 Nov 27. PMID 19945857
- [Result] Brandes AA, Stupp R, Hau P, et al.: EORTC Study 26041-22041: phase I/II study on concomitant and adjuvant temozolomide (TMZ) and radiotherapy (RT) with or without PTK787/ZK222584 (PTK/ZK) in newly diagnosed glioblastoma: results of a phase I trial. [Abstract] J Clin Oncol 25 (Suppl 18): A-2026, 2007.